CLINICAL TRIAL: NCT03962478
Title: Combined Stent Insertion and High-intensity Focused Ultrasound Ablation for Pancreatic Carcinoma With Biliary Obstruction
Brief Title: Combined Stent Insertion and HIFU Ablation for Pancreatic Carcinoma With Biliary Obstruction
Acronym: HIFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190522-021
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Pancreatic Carcinoma; Biliary Obstruction
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stent with high-intensity focused ultrasound ablation (Experimental): Patients undergo stent insertion with high-intensity focused ultrasound ablation on day 1.
  Interventions: Device: biliary stent and high-intensity focused ultrasound ablation system
- Stent without high-intensity focused ultrasound ablation (Active Comparator): Patients undergo stent insertion on day 1.
  Interventions: Device: biliary stent

INTERVENTIONS:
Device: biliary stent and high-intensity focused ultrasound ablation system — Self-expandable biliary nitinol alloys stent and YDME FEP-BY02 high-intensity focused ultrasound equipment
  Arms: Stent with high-intensity focused ultrasound ablation
Device: biliary stent — Self-expandable biliary nitinol alloys stent
  Arms: Stent without high-intensity focused ultrasound ablation

SUMMARY:
The purpose of this study is to compare the clinical effectiveness and long-term outcomes between patients with pancreatic carcinoma and biliary obstruction who are treated by stent insertion with or without high-intensity focused ultrasound ablation.

DETAILED DESCRIPTION:
Distal malignant biliary obstruction is a common problem in patients with pancreatic carcinoma. In unresectable pancreatic carcinomas, percutaneous stent placement has been pivotal in providing relief from obstructive jaundice, improving the quality of life, and allowing the maintenance of anticancer treatment.

Venous chemotherapy, transcatheter arterial chemoembolization, or radiotherapy have been used to prolong stent patency and survival after stent insertion for patients with pancreatic carcinoma and biliary obstruction. High-intensity focused ultrasound ablation is a noninvasive and atoxic treatment of malignant tumor using focused ultrasound energy from an extracorporeal source that is targeted within the body resulting in thermally induced necrosis and apoptosis.

The purpose of this study is to compare the clinical effectiveness and long-term outcomes between patients with pancreatic carcinoma and biliary obstruction who are treated by stent insertion with or without high-intensity focused ultrasound ablation.

ELIGIBILITY:
Inclusion Criteria:

1. malignant distal biliary obstruction;
2. pathologically diagnosed pancreatic carcinoma;
3. unresectable cases.

Exclusion Criteria:

1. inability to obtain informed consent;
2. Eastern Cooperative Oncology Group performance status of 4;
3. life expectancy of 3 months or less;
4. biliary obstruction that was not directly caused by pancreatic carcinoma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2020-02-08 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
6-month survival rate | From the date of randomization until the date of first documented death from any cause, assessed up to 12 months
  From the date of randomization until the date of first documented death from any cause.

SECONDARY OUTCOMES:
Stent patency | From the date of randomization until the date of first documented stent dysfunction, assessed up to 10 months
  Stent dysfunction is suspected when the patient experiences recurrence of jaundice.
Stent dysfunction free survival | From the date of randomization until the date of first documented stent dysfunction or the date of death from any cause, whichever came first, assessed up to 10 months.
  From the date of randomization until the date of first documented stent dysfunction or the date of death from any cause, whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Cao, MD, Principal Investigator — Xuzhou Central Hospital
Locations (1):
- Xuzhou Central Hospital, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.

REFERENCES:
- [Background] Niu S, Cheng L, Qiao Y, Fu YF, Cao C. Combined Stent Insertion and High-intensity Focused Ultrasound Ablation for Patients With Malignant Obstructive Jaundice. Surg Laparosc Endosc Percutan Tech. 2016 Dec;26(6):488-492. doi: 10.1097/SLE.0000000000000327. PMID 27783026
- [Derived] Zhang FQ, Li L, Huang PC, Xia FF, Zhu L, Cao C. Stent Insertion With High Intensity-Focused Ultrasound Ablation for Biliary Obstruction Caused by Pancreatic Carcinoma: A Randomized Controlled Trial. Surg Laparosc Endosc Percutan Tech. 2021 Feb 17;31(3):298-303. doi: 10.1097/SLE.0000000000000918. PMID 33605677